CLINICAL TRIAL: NCT04794634
Title: Relationship Between Alzheimer Disease and Diminution of the Three Macular Nervous Retinal Layers
Acronym: RETEVAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2021_843_0006
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Optical Coherence Tomography; Optical Coherence Tomography Angiography; Retinal Thickening; Alzheimer Disease; Lewy Body Disease; Retina; Cortical Atrophy; Retinal Nerve Fibres Layer
Keywords: Optical coherence tomography; Optical coherence tomography angiography; Retinal Thickening; Alzheimer Disease; Lewy Body Disease; Retina; Cortical Atrophy; Retinal Nerve Fibres Layer; Cell Ganglion Layer; Intern Plexiform Layer
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alzheimer Disease (Experimental)
  Interventions: Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Optical coherence tomograpohy angiography (OCTA)
- Lewy body disease (Experimental)
  Interventions: Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Optical coherence tomograpohy angiography (OCTA)
- healthy patient (Active Comparator)
  Interventions: Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Optical coherence tomograpohy angiography (OCTA)

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography (OCT) — to make a complete ophthalmological and neurological examination, an OCT to AD and to compare their results with LD and controls subjects
Diagnostic Test: Optical coherence tomograpohy angiography (OCTA) — to make a complete ophthalmological and neurological examination, an OCT and OCTA, to AD and to compare their results with LD and controls subjects

SUMMARY:
Alzheimer disease is hard, long and expensive to diagnose. In order to help the clinician, a new biomarker in Alzheimer disease seems to be very useful. The retina, as a window of the brain, could offer a new way to diagnose this common disease. Indeed, a retinal atrophy could especially appear in Alzheimer disease. Besides, many aspects about retinal alteration, visual function and their link with the disease deserve to be more explored. So as to fill these gaps, a new study about retinal specificity in Alzheimer disease appears to be relevant.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a consultation in the Research and Resources Memory Center of Amiens (RRMC) ,
* patients registered in the Alzheimer National Bank and having an Alzheimer Disease based on NIA-AA (McKahnn2011)and IWG2 (Dubois et al, 2014) criteria or, having a Lewy body disease based on revised criteria of McKeith et al 2020
* patients having a complete neuropsychological evaluation including a visual inspection time.
* patients having a MMSE ≥ 18/30 so as to ensure a good homogeneity of the group and to have an adequate ocular exam's quality.
* patients having an available MRI in the CHU's database including a 3DT1 sequence
* patients having a visual acuity better than 5/10, spherical refraction of +/- 5D, an astigmatism < 3D and an applanation IOP <22mmHg

Exclusion Criteria:

* Any other neurocognitive disorder
* Any other optical neuropathy including glaucoma
* All kind of retinal disease (diabetic retinopathy, age-related macular degeneration…)
* Diabetes mellitus
* Uncontrolled hypertension blood pressure
* Any ophthalmological conditions interfering with a good ocular examination or OCT quality (cataract, corneal opacity..)
* Severe dementia preventing a good ophthalmological examination
* Not consenting patient
* Patient with guardianship or curatorship having symptoms preventing a good ophthalmological examination (agitation, unstable ocular fixation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Variation of retinal nerve fibres layer (RNFL) thickness in AD patient compared to healthy and LMD patients | one day
  Thickness of retinal nerve fibres layer (RNFL), ganglion cell layer (CGL), intern plexiform layer (IPL) within the macular zone of patients suffering from AD.
Variation of ganglion cell layer (CGL) thickness in AD patient compared to healthy and LMD patients | one day
  Thickness of retinal nerve fibres layer (RNFL), ganglion cell layer (CGL), intern plexiform layer (IPL) within the macular zone of patients suffering from AD.
Variation of intern plexiform layer (IPL) thickness in AD patient compared to healthy and LMD patients | one day
  Thickness of retinal nerve fibres layer (RNFL), ganglion cell layer (CGL), intern plexiform layer (IPL) within the macular zone of patients suffering from AD.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No